CLINICAL TRIAL: NCT05060289
Title: A Prognostic Model for Drug-induced Liver Injury in China : A Multi-center, Prospective Cohort Study
Brief Title: A Prognostic Model for Drug-induced Liver Injury in China
Acronym: DILI-PM
Status: Recruiting | Type: Observational
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhao Xinyan, Professor, Beijing Friendship Hospital
Other Study IDs: 2021-P2-290-01
Record Dates: First submitted 2021-09-14; First posted 2021-09-29 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-01

CONDITIONS: Drug-induced Liver Injury
Keywords: prognostic model(s); biomarker(s); endpoint event(s)
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — serum, plasma, liver histopathology (if any)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Modeling group: The data of modeling group is used to construct a predictive model of DILI endpoint events.
- Validation group: Validation group is used to validate the predictive model externally.

SUMMARY:
A prospective, multi-center, non-interventional cohort study is going to conduct to explore the clinical characteristics, culprit drug(s) or herb(s), outcomes and risk factors of Drug-induced liver injury (DILI) in China and screen novel serum markers.

A prognostic model incorporating with the novel serum marker(s) for DILI would be established and validated to imporve the prognosis of patients in China .

DETAILED DESCRIPTION:
Research Objectives:

1. To establish a standardized multi-center, prospective DILI cohort nationwide and obtain long-term prognostic data.
2. To establish and verify prognostic model(s) of DILI in China.
3. To explore novel serum biomarkers for the prognosis of DILI.

ELIGIBILITY:
Inclusion Criteria:

1. RUCAM ≥6 and met one of the following biochemical conditions: (1) ALT≥5 ULN, (2) or ALP ≥2 ULN, (3) or ALT≥3 ULN and TBil≥2 ULN.
2. RUCAM between 3-5, five experienced hepatologists in leading site evaluate and vote the diagnosis of DILI, the case would be enrolled if only ≥4 out of 5 hepatologists agree with the diagnosis.
3. Onset to enrollment ≤3 months.

Exclusion Criteria:

1. Hepatotropic viral infection: hepatitis A, B, C, D and E.
2. Non-hepatotropic viral infection: cytomegalovirus (CMV) and Epstein-Barr virus (EBV), etc.
3. Hypoxic ischemic hepatitis and congestive liver disease.
4. Alcohol consumption: male >40g/d, female >20g/d, and ≥5 years.
5. Biliary obstruction, primary biliary cholangitis; primary sclerosing cholangitis.
6. Autoimmune hepatitis: International Autoimmune Hepatitis Group (IAHG) simplified score ≥6 or complicated score ≥10, or differentiation from autoimmune hepatitis is impossible during enrollment.
7. Parasitic infection.
8. Sepsis.
9. Previous liver transplantation or bone marrow transplantation.
10. Pregnancy or lactation.
11. Genetic and metabolic liver diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult with drug-induced liver injury
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
death/liver transplantation | 1 year
  DILI has a primary, contributory role for the death (liver-related mortality) or no role for the death (all-cause mortality) .
  DILI is the primary indication for liver transplantation.
acute liver failure | 1 year
  Acute liver failure is defined as elevated bilirubin and prolonged international normalized ratio (INR) ≥1.5 accompanied by mental disturbance within 26 weeks after DILI onset without underlying chronic liver diseases.

SECONDARY OUTCOMES:
chronic DILI | 2 years
  Chronicity is defined as the presence of any one of the following: (i) persistently elevated liver biochemistry indexes; (ii) radiological or histological evidence of persistent liver injury at one year after DILI onset.
recovery | 2 years
  Recovery status is defined as clinical and biochemical resolution within 1 year after DILI onset, with alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤40 U/L, alkaline phosphatase (ALP) ≤150 U/L, and total bilirubin (TB) ≤1.5 upper limits of normal (ULN) (25.65 μmol/L).

CONTACTS AND LOCATIONS:
Overall Officials: Xinyan Zhao, Study Chair — Beijing Friendship Hospital; Zhengsheng Zou, Principal Investigator — Beijing 302 Hospital; Yu Chen, Principal Investigator — Beijing You 'an Hospital, Capital Medical University; Juan Li, Principal Investigator — Qinghai People's Hospital; Pingying Li, Principal Investigator — Qinghai People's Hospital; Xiaoju Liu, Principal Investigator — Qinzhou First People's Hospital; Liang Wang, Principal Investigator — Lanzhou University Second Hospital; Juan Luo, Principal Investigator — Hebei CNPC Central Hospital; Huahua Wang, Principal Investigator — Jiaozuo People's Hospital; Hui Wang, Principal Investigator — Jiaozuo People's Hospital; Jikang Yang, Principal Investigator — Jiaozuo People's Hospital; Doudou Hu, Principal Investigator — Qingdao Municipal Hospital; Qiuju Tian, Principal Investigator — The Affiliated Hospital of Qingdao University; Rongkuan Li, Principal Investigator — The Second Affiliated Hospital of Dalian Medical University; Lu Li, Principal Investigator — Peking University Third Hospital; Liuyi Chang, Principal Investigator — Yuncheng Central Hospital; Lu Zhang, Principal Investigator — Beijing Ditan Hospital; Yuanjiao Gao, Principal Investigator — Beijing Ditan Hospital
Locations (13):
- China (13):
  - Beijing 302 Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing
  - Beijing You 'an Hospital, Capital Medical University, Beijing
  - Beijing Ditan Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - The Second Affiliated Hospital of Dalian Medical University, Dalian
  - Qinzhou First People's Hospital, Guangxi
  - Hebei CNPC Central Hospital, Hebei
  - Jiaozuo People's Hospital, Jiaozuo
  - The Second Hospital of Lanzhou University, Lanzhou
  - The Affiliated Hospital of Qingdao University, Qingdao
  - Qinghai People's Hospital, Qinghai
  - Yuncheng Central Hospital, Yuncheng

IPD SHARING:
Plan to Share IPD: No